CLINICAL TRIAL: NCT00874809
Title: A Pilot Study to Explore Basal Insulin Dosing Requirements in Patients With Type 2 Diabetes Treated With Insulin Pump Therapy
Brief Title: Diabetes Mellitus Type 2 Basal Insulin Dosing Requirements Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Care Center (Industry)
Collaborators: Animas Corporation (Industry)
Responsible Party: Principal Investigator, Allen B. King, MD, Principal Investigator, Diabetes Care Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1799
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin pump; DM Type 2; CGMS; basal rate
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin Treatment (Other): There is only one arm for this study using lispro insulin administered by insulin pump.
  Interventions: Device: CGMS with an insulin pump using rapid acting insulin

INTERVENTIONS:
Device: CGMS with an insulin pump using rapid acting insulin — To determine basal changes subject will wear a CGMS with an insulin pump infusing rapid acting insulin
  Other Names: Continuous Glucose Monitoring System (CGMS)

SUMMARY:
The main purpose of this study is to determine the number of daily basal insulin rate changes that are needed to achieve short-term near normal glucose control in insulin pump patients with type 2 diabetes

DETAILED DESCRIPTION:
Subjects will be taught CHO counting after which they will be introduced to an insulin pump. They will wear the insulin pump for three weeks to adjust to the pump and its functions. Then the subject will wear a Continuous Glucose Monitoring System to determine rate changes needed to achieve short-term near normal glucose control. The primary endpoint is what are the mean number of changes in the basal infusion rate and what are the mean differences and mean duration of these changes. The secondary endpoint is what mathematical formulas describe the relationship between the dosing factors and do they significantly differ from those previously established by King and Armstrong.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes > 3month duration
* Age 18
* Hb A1C <12%
* On any hypoglycemic therapy including insulin for 5 patients and 5 patients naive to insulin and failing oral treatment
* Normal creatine
* Negative for GAD antibodies
* SMBG >4/d and willing/able to comply with study requirements
* Demonstrated adherence to visits and instructions.

Exclusion Criteria

* Severe hypoglycemic during the last month
* Severe cardiac, pulmonary or cerebral disease
* Demonstrated non compliance with clinical recommendations
* Pregnancy, nursing or women who could potentially become pregnant
* Presence of physical, psychological or cognitive impairments that would interfere with adherence to an intensive insulin therapy program or compliance with dietary, diary keeping or maintenance of CGM sensor or pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
What are the mean number of changes in the basal infusion rate(change is defined as any alternation in the basal rate >0.1 U/hr) and what are the mean differences and mean duration (hrs) of these changes. | week six of study

SECONDARY OUTCOMES:
What mathematical formulas describe the relationship between the dosing factors and do they significantly differ from those previously established by King and Armstrong | week 6 of study

CONTACTS AND LOCATIONS:
Overall Officials: Allen B King, MD, Principal Investigator — Diabetes Care Center
Locations (1):
- Diabetes Care Center, Salinas, California, United States